CLINICAL TRIAL: NCT06252298
Title: A Phase I Clinical Study Evaluating the Safety and Efficacy of SCTC21C in Participants With CD38+ Hematologic Malignancies
Brief Title: A Clinical Study of SCTC21C in Participants With CD38+ Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCTC21C-X101
Record Dates: First submitted 2024-01-31; First posted 2024-02-09 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-01

CONDITIONS: Relapsed or Refractory Hematologic Malignancies
MeSH Terms: conditions — Recurrence; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose-finding and dose-expansion (Experimental): Dose-finding stage: The dose escalation in this study is pre-defined in nine dose groups. The dose escalation starts with 0.01mg and proceeds from low to high doses.
  Dose-expansion stage: Patients will be randomly assigned to receive different doses of SCTC21C at a ratio of 1:1. Doses of SCTC21C will be determined based on the data obtained in the Dose-finding stage.
  Interventions: Biological: SCTC21C

INTERVENTIONS:
Biological: SCTC21C — SCTC21C is injected to the participants subcutaneously and is tentatively scheduled to be administered weekly for the first two cycles, once every 2weeks for cycle3-6, and once every 4 weeks thereafter until the occurrence of progressive disease

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of SCTC21C in patients with CD38+ hematologic malignancies

DETAILED DESCRIPTION:
This is a multicenter, open-label, phase I study aimed to evaluate the safety, tolerability, pharmacokinetics（PK）, Pharmacodynamics（PD）, preliminary anti-tumor activity and immunogenicity of SCTC21C in patients with relapsed or refractory CD38+ hematologic malignancies.The study includes Dose-finding stage and Dose-expansion stage. In Dose-finding stage, participants will be assigned to receive sequentially higher doses of SCTC21C ranging from 0.01 to 960mg. In Dose-expansion stage, total of at least 20 participants will be randomly assigned to receive two different doses of SCTC21C at a ratio of 1:1.All participants will receive the treatment until disease progression or unacceptable drug-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 18 years old when signing ICF, weight ≥ 40 kg, ≤ 90 kg
2. Relapsed or refractory CD38+（confirmed by immunohistochemistry or flow cytometry） hematologic malignancies
3. Standard therapies failed or are unavailable or intolerant
4. Participants have at least one of the measurable lesions
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
6. Life expectancy ≥3 months
7. Participants with basically normal liver, kidney and heart functions
8. Hematology requirements: platelet≥75x10^9 /L,absolute neutrophil counts ≥ 1.0x10^9 /L, hemoglobin ≥ 8.0 g/dL
9. Women of childbearing potential (must have a negative blood pregnancy test within 7 days before the first dose) or male participants must use a highly effective method of contraception from signed ICF to 5 months after the last dose.All participants are prohibited from donating sperms or ova during the study period and 5 months after the last dose

Exclusion Criteria:

1. A history of allergic reactions to any SCTC21C injection or any excipients, or Participants with a history of severe drug allergy
2. Participants who have other antineoplastic drug (except hormones) or radiotherapy within four weeks prior to the first dose of study drug, or the participants who have received immunotherapy or anti-CD38 monoclonal antibody within 6 months
3. Adverse events from the previous treatment have not resolved to ≤ Grade 1
4. Participants with prior immunotherapy and Grade ≥ 3 cytokine release syndrome(CRS)
5. Central nervous system involvement
6. Participants with positive Human immunodeficiency virus (HIV) antibody
7. HBsAg positive with HBV-DNA titer higher than the lower limit of the test value of the research center, or HCV antibody positive with HCV-RNA titer higher than the lower limit of the test value of the research center
8. Active infections that require systemic treatment within 1 week prior to the first dose
9. History of additional malignant tumor or active autoimmune diseases,or participants with other serious medical conditions
10. Participants underwent major surgery within 4 weeks prior to the first dose, or had a surgical schedule during the study period
11. History of allogeneic hematopoietic stem cell transplantation or solid organ transplantation,or history of autologous hematopoietic stem cell transplantation within 6 months prior to screening
12. Participants with significant digestive system dysfunction that may affect drug intake, transport and absorption
13. Participants who have received live vaccines within 30 days prior to the first dose of study drug
14. Participants with mental disorders or poor compliance
15. Female participants who are breastfeeding
16. The Investigator determined that the participant is ineligible for the study for other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-08-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) and serious adverse event (SAE) | From the initiation of the first dose to the 45 days after the last dose
  To identify the incidence of TEAEs and SAE
The incidence of dose limiting toxicities （dose-finding stage） | Cycle 1 (28 days)
  To identify the DLTs

SECONDARY OUTCOMES:
Objective response rate (ORR) | Throughout the study treatment,an average of 1 year
  ORR is defined as the proportion of patients who have an objective remission

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chaoyang Hospital ,Capital Medical University, Beijing, Beijing Municipality, China